CLINICAL TRIAL: NCT01093001
Title: The Effect of Cardiac Pacing Leads on Tricuspid Regurgitation
Brief Title: Tricuspid Regurgitation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Yong-Mei Cha, Cardiovascular Division, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08-008690
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Tricuspid Regurgitation; Right Ventricular Dysfunction; Left Ventricular Dysfunction
Keywords: Reduce Tricuspid Regurgitation; Reduce Right Ventricular pacing; Lead position; Lead size
MeSH Terms: conditions — Tricuspid Valve Insufficiency; Ventricular Dysfunction, Right; Ventricular Dysfunction, Left | interventions — Caves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Lead size (Active Comparator): The pacemaker lead will be < or = to 7Fr. The ICD lead will be 9 Fr.
  Interventions: Other: Echo
- RV Lead position (Active Comparator): 50 patients will be randomized to RV apex lead placement.
  Interventions: Other: Echo
- Mid-Septum Lead position (Active Comparator): 50 patients will be randomized to RV mid-septum lead placement.
  Interventions: Other: Echo
- CS lead position (Active Comparator): 50 patients will have lead placed in the CS
  Interventions: Other: Echo

INTERVENTIONS:
Other: Echo — Two dimensional echocardiography will be performed to reassess Tricuspid Regurgitation.
  Arms: Lead size
Other: Echo — Two dimensional echocardiography will be performed to reassess Tricuspid Regurgitation
  Arms: RV Lead position
Other: Echo — Two dimensional echocardiography will be performed to reassess Tricuspid Regurgitation.
  Arms: Mid-Septum Lead position
Other: Echo — Two dimensional echocardiography will be performed to reassess Tricuspid Regurgitation.
  Other Names: Medtronic Starfix lead
  Arms: CS lead position

SUMMARY:
The effect of cardiac pacing leads on tricuspid regurgitation is unclear. This study will determine whether using a smaller diameter leads and an alternate position in the ventricle, the proximal septum, will reduce tricuspid regurgitation than larger leads placed in the apex.

DETAILED DESCRIPTION:
Leads are commonly placed in the right ventricular apex. It is not known whether placing similar leads higher on the septum where there will be less redundancy or pressure on the septal leaflet will change the extent and severity of tricuspid regurgitation following pacemaker/ICD implantation. Data has shown that right ventricular pacing can give rise to right ventricular dysfunction, which in turn may give rise to enlargement of the right ventricle and cause tricuspid regurgitation.

The study will answer the clinically relevant questions on device lead-related tricuspid regurgitation.

This study is a single center prospective study at the Mayo Clinic, Rochester. The study will enroll 200 eligible subjects and follow for 12 months. 50 pacemaker subjects will be randomized to right ventricular apex pacing 50 pacemaker subjects will be randomized to right ventricular septum pacing 50 pacemaker subjects will be randomized to left ventricular pacing via coronary sinus 50 ICD subjects will be enrolled with right ventricular apex pacing.

A baseline heart failure assessment and Two Dimensional echocardiography will be performed before device implant.

A Two Dimensional echo will be performed 24 hours after device implant. If significance TR is present a Three Dimensional echo will be performed. At 12 months post implant heart failure assessment and Two Dimensional echo will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of either sex

  * Patient is recommended to receive a pacemaker or an ICD
  * Provide informed consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* Congenital heart disease
* Pre-existing moderate or severe TR
* An existing pacemaker or defibrillator
* Pulmonary hypertension
* Pacemaker dependence
* Unable to give informed consent
* Not feasible for patient to be followed up at Mayo Clinic
* Acute myocardial infarction within 7 days

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2010-05; Primary Completion 2015-09 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Decrease in Tricuspid Regurgitation using smaller diameter lead and placing the lead on the proximal septum. | 12 months

SECONDARY OUTCOMES:
Left Ventricular lead placement will be associated with least amount of TR because of avoiding crossing the tricuspid valve and by virtue of relatively more synchronous ventricular contractions. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Mei Cha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] 1. Lin G, Nishimura R, Connolly H, Dearani J, Sundt T, Hayes D: Severe symptomatic tricuspid valve regurgitation due to permanent pacemaker or implantable cardioverter-defibrillator leads. JACC 2005; 45:1672-1675. 2. Leibowitz D, Rosenheck S, Pollak A, Geist M, Gilon D: Transvenous pacemaker leads do not worsen tricuspid regurgitation: a prospective echocardiographic study. Arrhythmias, Electrophysiology and Electrocardiography 2000; 93:74-77. 3. Kucukarslan N, Kirilmaz A, Ulusoy E, Yokusoglu M, Gramatnikovski N, Ozal E, Tatar H: Tricuspid insufficiency does not increase early after permanent implantation of pacemaker leads. J Card Surg 2006; 21:391-394. 4. Wilkoff B, Invesigators DT: The dual chamber and WI implantable defibrillator (DAVID) Trial: rationale, design, results, clinical implications and lessons for future trials. Cardiac Electrophysiol Review 2004; 7:468-472.